CLINICAL TRIAL: NCT05449470
Title: Alerting on Adverse Drug Reactions: Falls Prevention Improvement Through Developing a Computerized Clinical Support System: Effectiveness of Individualized medicaTion Withdrawal
Brief Title: A Clinical Decision Support System and Patient Portal for Preventing Medication-related Falls in Older Patients
Acronym: ADFICE_IT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: VU University of Amsterdam (Other)
Responsible Party: Principal Investigator, Prof. dr. Nathalie van der Velde, Full Professor Geriatric medicine (internal medicine), Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021_061
Record Dates: First submitted 2022-03-24; First posted 2022-07-08 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Fall; Fall Injury; Fall Patients; Accidental Fall; Deprescriptions; Polypharmacy; Aged; Aged, 80 and Over
Keywords: fall prevention; fall-risk increasing drugs (FRIDs); older out-clinic patients; injurious falls; prediction model; clinical decision support system; patient portal; Shared Decision Making (SDM); medication withdrawal
MeSH Terms: interventions — Patient Portals

STUDY DESIGN:
Intervention Model Description: Patients (in both arms) who schedule an appointment will receive a letter containing information on the objectives and procedures of the study and an invitation to participate. For patients in the intervention arm, the invitation letter will also include a printed QPL and a link to the Patient portal. At this point, the Patient portal will only provide information on their upcoming visit as well as educational material regarding falls prevention.
  At the falls clinic the assessments will be carried out as usual. In the intervention group, the physician will use the CDSS during the consultation. Consultations in the control group are carried out as usual. After the consultation, patients and their caregivers (if applicable) will be asked to fill out a set of questionnaires. After the visit to the falls clinic, patients in the intervention group will be able to review their consultation with the physician and their estimated fall risk in the patient portal.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CDSS and patient portal (Experimental): The intervention includes the combined use of the clinical decision support system (CDSS) that provides deprescribing advice and a personalized risk prediction and a patient portal.
  Interventions: Device: CDSS; Device: Patient Portal
- Care as usual (No Intervention): Care as usual

INTERVENTIONS:
Device: CDSS — A clinical decision support system (CDSS) that provides deprescribing advice and a personalized risk prediction
  Other Names: Clinical Decision Support System
  Arms: CDSS and patient portal
Device: Patient Portal — A Patient Portal that helps patients prepare for their fall clinic visit by giving them information about falls, falls prevention, and medication-related falls. After the fall clinic visit, the Patient Portal also shows the personalized fall-risk and treatment advice.
  Other Names: Valportaal
  Arms: CDSS and patient portal

SUMMARY:
Falls in older adults represents a growing public health challenge. The use of certain medication is recognized as an important modifiable risk factor for falls. Research indicates fall-risk increasing drug (FRID) deprescribing is effective in reducing falls but difficult to initiate and to sustain over longer periods of follow-up. A clinical decision support system (CDSS) and patient portal for communicating medication-related fall risk to fall clinic patients may improve joint medication management between patients and physicians and consequently reduce the incidence of injurious falls.

DETAILED DESCRIPTION:
This study investigates the effectiveness and cost-effectiveness of the concurrent use of a CDSS and a patient portal for personalized FRID deprescribing, and will be assessed through a multicenter cluster-randomized controlled trial among new fall clinic patients, aged 65 years or older. The main study parameter is the time to first injurious fall. The primary objective of the ADFICE_IT study is to investigate the effects of a CDSS and accompanying patient portal for optimizing FRID deprescribing on injurious falls. This study has three secondary objectives. First, the effect of the CDSS and patient portal on a number of secondary outcomes will be investigated. Second, a process evaluation to evaluate the implementation of the CDSS and patient portal will be conducted. Third, the cost-effectiveness of the CDSS and patient portal will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* History of at least one fall in the past year;
* A Mini-Mental State Examination (MMSE) score of 21 points or higher or equivalently a Montreal Cognitive Assessment (MOCA) Dutch score of 16 points or higher;
* Use of at least one fall-risk increasing drug (FRID); and
* Sufficient command of the Dutch language in speech and writing.

Exclusion Criteria:

* Active participation in another study;
* Life expectancy of less than one year: and/or
* Suffering from severe mobility impairment (i.e. bedridden, e.g. inability to walk short distances with assistance of a walking aid).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2022-07-07 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Time to first injurious fall | 12 months
  This concerns the time to the first injurious fall. An injurious fall is defined as a fall resulting in wounds, bruises, sprains, cuts, medically recorded fractures, head or internal injury, requiring medical/health professional examination, accident and emergency treatment, or inpatient treatment.

SECONDARY OUTCOMES:
Number of injurious falls | 12 months
  This concerns the total number of injuirous falls over the course of 12 months. An injurious fall is defined as a fall resulting in wounds, bruises, sprains, cuts, medically recorded fractures, head or internal injury, requiring medical/health professional examination, accident and emergency treatment, or inpatient treatment.
Total number of falls | 12 months
  Total number of any fall (I.e. a fall that results in no injuries, or minor, moderate, or severe injuries)
Time to first fall resulting in any injuries | 12 months
  I.e. a fall that results in minor, moderate, or severe injuries
Total number of falls resulting in any injuries | 12 months
  I.e. a fall that results in minor, moderate, or severe injuries
Time to first non-injurious fall | 12 months
  I.e. a fall that results in no injuries
EuroQol-5D-5L (EQ-5D-5L) | at baseline, 3 months, 6 months, and 12 months
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension in the EQ-5D-5L has five response levels: no problems (Level 1); slight; moderate; severe; and extreme problems (Level 5). Furthermore, it includes a visual analogue scale (EQ-VAS) which provides a single global rating of self-perceived health and is scored on a 0 (worst health imaginable) to 100 (best health imaginable) scale.
The Older Persons and Informal Caregivers Minimum Data Set-Short Form (TOPICS-SF) | at baseline and 12 months
  Data as measured by the The Older Persons and Informal Caregivers Minimum Data Set-Short Form (TOPICS-SF) will be analysed based on the preference-weighted score, ranging from 1.90 to 9.78, with higher scores reflecting a better health status, as perceived by the respondent. The TOPICS - Short Form 2017 including Casemix forms were developed in collaboration with the Nederlandse Vereniging voor Klinische Geriatrie (NvKG - Dutch Association for Clinical Geriatrics) to use as a Patient Reported Outcome Measure (PROM) in the Dutch outpatient and clinical daily practice.
iMTA Productivity Cost Questionnaire (iPCQ) | at baseline, 3 months, 6 months, and 12 months
  Direct and indirect costs related to the intervention and care as usual will be assessed using the iMTA Productivity Cost Questionnaire (iPCQ).
iMTA Medical Consumption Questionnaire (iMCQ) | at baseline, 3 months, 6 months, and 12 months
  The iMTA Medical Consumption Questionnaire (iMCQ) is an instrument for measuring medical consumption. The iMCQ includes questions related to frequently occurring contacts with health care providers.

OTHER OUTCOMES:
Feasibility assessed by number of CDSS and patient portal use | 12 months
  To assess the feasibility of the intervention, the investigators will use data logged by the CDSS and patient portal to understand how (often) the CDSS and patient portal are used
Percentage of physicians attending the CDSS training via a questionnaire | 12 months
  To assess the feasibility of the intervention, the investigators will look at the percentage of physicians who attended the CDSS training. More specifically, this will be measured by asking physicians whether they attended the CDSS training online, offline or not at all as part of the CDSS user satisfaction questionnaire.
Correlation of percentage of physicians attending the CDSS training and CDSS user satisfaction | 12 months
  The correlation between the proportion of a department's staff members who did/did not participate in the CDSS training and user satisfaction regarding the CDSS will be assessed.
CDSS user satisfaction | 12 months
  To assess the feasibility of the intervention, the investigators will study the satisfaction regarding the CDSS (i.e. physician evaluations of the CDSS). Agreement with satisfaction statements will be scored on a 7-point Likert scale (1= totally disagree; 7 = totally agree).
Technology Acceptance Model (TAM) | at baseline
  The Technology Acceptance Model (TAM) is designed to measure the adoption of a new technology/system based on user attitudes. 6 items aim to measure Perceived Usefulness on a 7-point Likert scale (1=totally disagree; 7 = totally agree), and 6 items aim to measure Perceived Ease of Use on a 7-point Likert scale (1=totally disagree; 7 = totally agree). Intention to use is measured through 1 item on a 7-point Likert scale (1=totally disagree; 7 = totally agree)
Website Satisfaction Scale (WSS) | at 3 months
  The Website Satisfaction Scale (WSS) measures satisfaction with comprehensibility, satisfaction with attractiveness, and satisfaction with emotional support through 12 items, for each sub scale using a 7-point Likert response scale, ranging from 1 'totally disagree' to 7 'totally agree'.
Observer OPTION Multiple Chronic Conditions (OPTION-MCC) | 12 months
  Videotaped consultations will be coded on triadic decision making in older patients with multiple chronic conditions by using the Observer OPTION Multiple Chronic Conditions (OPTION-MCC) coding scheme. Six types of physicians', patients', and caregivers' behaviors are coded. Physicians' behavior is coded on a 5-point scale (0= The behavior is not observed; 4=The behavior is executed to a very high standard), patients' behavior is coded on a 3-point scale (0=No or minimal participation, e.g. only yes or no; 2=Active participation, answers questions and asks questions, brings in own ideas and shares perceptions), and informal caregivers' behavior is coded on a 3-point scale (0=No or minimal participation, e.g. only yes or no; 2=Active participation, answers questions and asks questions, brings in own ideas and shares perceptions)
Rate of adherence to new medication plan using pharmacy records | 12 months
  To assess adherence to the medication advice, the investigators will compare a patient's new medication advice with their pharmacy records to determine whether a patient adheres to the new medication advice or whether they (eventually) change back to their old medication
Number of falls calendar entries | 12 months
  To assess adherence to the medication advice, the investigators will compare the new medication advice with falls calender entries on medication use to determine whether a patient adheres to the new medication advice or whether they (eventually) change back to their old medication
iSHARE | 12 months
  To evaluate how the intervention facilitates SDM, the investigators will use the iSHAREpatient and iSHAREphysician questionnaires. The iSHAREphysician consists of 16 items scored on a 6-point Likert scale (1= did not do this at all; 6 = completely did this). The iSHAREpatient consists of 16 items scored on a 6-point Likert scale (1= did not do this at all; 6 = completely did this). Dimension scores (range, 0-5) and a total score (the sum of the dimension scores; range, 0-30) for both iSHARE questionnaires will be calculated. The investigators will then apply a linear transformation to obtain a 0 to 100 total score ((score/30)*100). Higher dimension and total scores indicate higher levels of SDM.
Decisional Conflict Scale (DCS; low literacy scale) | at baseline
  To evaluate how the intervention facilitates SDM, the investigators will use the Decisional Conflict Scale (DCS; low literacy scale). This scale consists of 10 questions, scored on 3 response categories (yes, do not know, no).
Preparation for Decision-making scale (PrepDM) | at baseline
  To evaluate how the intervention facilitates SDM, the investigators will use the Preparation for Decision-making scale (PrepDM). This scale consists of 10 items, scored on a 5-point Likert scale (1= not at all; 5 = a great deal)
Netherlands Patient Information Recall Questionnaire (NPIRQ) | 12 months
  To evaluate how the intervention facilitates SDM, the investigators will use the Netherlands Patient Information Recall Questionnaire (NPIRQ). This questionnaire consists of open questions.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie van der Velde, MD, PhD, Principal Investigator — Amsterdam UMC, Academic Medical Center, University of Amsterdam, Amsterdam, The Netherlands; Natasja M van Schoor, PhD, Principal Investigator — Amsterdam UMC, Vrije Universiteit Amsterdam, Amsterdam Public Health, Amsterdam, the Netherlands; Annemiek J Linn, PhD, Study Director — Amsterdam School of Communication Research, University of Amsterdam, Amsterdam, The Netherlands
Locations (10):
- Netherlands (10):
  - Radboud universitair medisch centrum, Nijmegen, Gelderland
  - Elisabeth-TweeSteden Ziekenhuis, Tilburg, North Brabant
  - Ziekenhuis Amstelland, Amstelveen, North Holland
  - Amsterdam UMC, locatie VUmc, Amsterdam, North Holland
  - OLVG, Amsterdam, North Holland
  - Amsterdam UMC, locatie AMC, Amsterdam, North Holland
  - Spaarne Gasthuis, Haarlem, North Holland
  - Medisch Centrum Leeuwarden, Leeuwarden, Provincie Friesland
  - UMC Groningen, Groningen
  - St. Antonius Ziekenhuis, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided
Currently no plan

REFERENCES:
- [Derived] Groos SS, de Wildt KK, van de Loo B, Linn AJ, Medlock S, Shaw KM, Herman EK, Seppala LJ, Ploegmakers KJ, van Schoor NM, van Weert JCM, van der Velde N. Development of the ADFICE_IT clinical decision support system to assist deprescribing of fall-risk increasing drugs: A user-centered design approach. PLoS One. 2024 Sep 5;19(9):e0297703. doi: 10.1371/journal.pone.0297703. eCollection 2024. PMID 39236057
- [Derived] de Wildt KK, van de Loo B, Linn AJ, Medlock SK, Groos SS, Ploegmakers KJ, Seppala LJ, Bosmans JE, Abu-Hanna A, van Weert JCM, van Schoor NM, van der Velde N; ADFICE_IT study team. Effects of a clinical decision support system and patient portal for preventing medication-related falls in older fallers: Protocol of a cluster randomized controlled trial with embedded process and economic evaluations (ADFICE_IT). PLoS One. 2023 Sep 26;18(9):e0289385. doi: 10.1371/journal.pone.0289385. eCollection 2023. PMID 37751429